CLINICAL TRIAL: NCT01040923
Title: Validation of the Cardiosond Sonospectrographic Digital Electronic Stethoscope in Diagnosing Coronary Artery Disease Versus CT Angiography
Brief Title: Comparison of Digital Electronic Stethoscope to Computed Tomography (CT) Angiography in Detection of Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: SonoMedica, Inc. (Industry)
Collaborators: North Shore University Hospital (Other); Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: SM-C102
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease
Keywords: CAD; Diagnostic
MeSH Terms: conditions — Coronary Artery Disease; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac CT: All patients in the study will be those presenting themselves for cardiac CT angiography who meet the proper inclusion / exclusion criteria
  Interventions: Device: CardioSond Cardiac Sonospectrographic Analyzer

INTERVENTIONS:
Device: CardioSond Cardiac Sonospectrographic Analyzer — The CardioSond is a completely noninvasive, FDA 510(k) cleared digital electronic stethoscope designed to detect heart sounds and murmurs using ultrasensitive acoustic technology.
  Other Names: CardioSond; CSA

SUMMARY:
The study is designed to evaluate the predictive diagnostic accuracy of SonoMedica's CardioSond digital electronic stethoscope in the detection of coronary artery disease (CAD) in patients without known disease who are referred to cardiac computed tomography angiography (CT scans).

DETAILED DESCRIPTION:
The CardioSond is a completely noninvasive medical device which detects heart sounds and murmurs using ultrasensitive acoustic technology. The CardioSond produces a flow micro bruit score which is used to determine the likelihood of coronary artery disease.

The CardioSond exam will be given to patients who agree to participate in the study upon signing of an informed consent form and prior to the administration of beta blocker agents and / or vasodilators as part of the normal cardiac CT angiography protocol.

CardioSond data will be sent to an independent acoustic core lab which will determine data quality and produce a flow micro bruit score. CT angiography data will be analyzed by staff at North Shore University Hospital.

A data review panel lead my the principal investigator will examine the results of both the CardioSond and CT angiography data to determine the accuracy of the CardioSond in detecting CAD in the study population at large and in specific patient subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are undergoing routine screening coronary CT angiography
* Willingness to sign informed consent form

Exclusion Criteria:

* Inability to provide informed consent form
* Age less than 21 years
* Any contraindications to coronary CT angiography
* Known atherosclerotic heart disease, including a history of prior myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery or an established diagnosis of CAD by prior X-ray or CT angiography
* Supraventricular or ventricular arrhythmias that would be expected to affect CT-angiography image quality (e.g., atrial fibrillation, atrial flutter, ventricular tachycardia, bigeminy, and trigeminy). Patients with isolated premature atrial contractions and premature ventricular contractions may enroll.
* Use of intravenous vasodilators
* Any pulmonary conditions that would create abnormal physical findings that would interfere with the fidelity of the cardiac sound recording (e.g., obstructive pulmonary disease, such as asthma or COPD, with audible wheezing).
* Presence of audible aortic or pulmonic diastolic murmurs, tricuspid or mitral flow diastolic murmurs, or continuous murmurs

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be sourced from patients presenting themselves for cardiac CT angiography who meet appropriate inclusion / exclusoin criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the CardioSond digital electronic stethoscope's flow micro bruit score as an indication of the probability of coronary artery disease in patients without know disease versus the results of cardiac CT angiography. | Post collection of CardioSond and CT angiography data

SECONDARY OUTCOMES:
Comparison of CardioSond's flow micro bruit score as an indication of the probability of coronary artery disease against the results of cardiac CT angiography in patient subgroups including age, sex, body mass index, location and severity of disease. | Upon collection of CardioSond and CT angiography data

CONTACTS AND LOCATIONS:
Overall Officials: Amgad N Makaryus, MD, Principal Investigator — North Shore University Hospital; Diane Dellilune, RN, Study Director — North Shore University Hospital
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States